CLINICAL TRIAL: NCT07058688
Title: A Multicenter, Randomized, Double-masked, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NTRX-07 in Subjects With Mild Cognitive Impairment or Mild to Moderate Alzheimer's Disease
Brief Title: A Study of NTRX-07 in Participants With Alzheimer's Disease
Acronym: SPPN-AD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroTherapia, Inc. (Industry)
Collaborators: Cruint Global Consulting Pte Ltd (Unknown); Firalis SA (Industry); Pharma-Regist Kft. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTRX-07-C201; 2024-517957-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-15; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: clinical pharmacology; neuroinflammation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neuroinflammatory Diseases

STUDY DESIGN:
Intervention Model Description: A randomized, double-masked, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- QD Dosing (Experimental): NTRX-07 90 mg as two 45 mg tablets administered orally once per day
  Interventions: Drug: NTRX-07
- Placebo (Placebo Comparator): Two tablets matching the Experimental treatment administered orally once per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTRX-07 — Orally administered CB2 agonist
  Other Names: MDA7
  Arms: QD Dosing
Drug: Placebo — Inactive matched comparator
  Arms: Placebo

SUMMARY:
1. Study Overview NeuroTherapia Inc. is conducting a clinical study to explore the safety and effects of a new drug called NTRX- 07. This drug targets people with mild cognitive impairment (MCI) or mild to moderate Alzheimer's disease (AD). The study's primary focus is on safety and how the drug interacts with the body over a short-term period of 28 days. This research is important as it aims to find new ways to manage symptoms and slow the progression of AD.
2. Key Objectives Primary Objective:

   * To assess the safety and tolerability of NTRX-07 in patients with AD.
   * Safety and tolerability will be measured by monitoring any side effects or adverse events in participants during and after the treatment period.

   Secondary Objective:
   * To study how NTRX-07 is processed by the body, including how it is absorbed, distributed, metabolized, and eliminated.
   * This includes measuring the drug levels in the blood and cerebrospinal fluid (CSF) over time.
3. Study Design • Type of Study:

   o A randomized, double-masked, placebo-controlled study. "Randomized" means participants are randomly assigned to receive either the actual drug (NTRX-07) or a placebo (an inactive substance). "Double-masked" indicates that neither the participants nor the researchers know who receives the real drug or the placebo, reducing bias and ensuring objective results.

   • Participants:
   * 48 individuals with MCI or mild to moderate AD.

     • Treatment Groups:
   * Participants will be split into two groups: 24 will receive NTRX-07, and 24 will receive a placebo.

     • Duration:
   * The study will last up to 7-10 weeks for each participant, including a 28-day period during which they take the drug or placebo daily.
4. Study Procedures

   • Screening Period:
   * Before starting the treatment, participants will undergo a screening period of up to 45 days. During this time, they will have tests to confirm their eligibility, including physical exams, blood tests, cognitive assessments, and brain imaging (MRI).

     • Treatment Period (28 days):
   * Participants will take the study drug or placebo daily for 28 days. During this period, they will visit the study center for evaluations, including safety checks, cognitive tests, blood and CSF sampling, and EEG tests (to measure brain activity).

     • Follow-Up:
   * After the treatment period, participants will have a follow-up visit 7 days later for final safety assessments.
5. Safety Monitoring and Assessments

   * The study's primary focus is on safety. Researchers will monitor participants closely for any adverse events, such as side effects, throughout the study.
   * Safety assessments will include monitoring vital signs (blood pressure, heart rate, temperature), conducting laboratory tests (blood and urine analysis), performing physical examinations, and using electrocardiograms (ECGs) to monitor heart health.
6. Exploratory Assessments

   • Although this study primarily focuses on safety, researchers will also conduct exploratory assessments to observe any potential positive effects of NTRX-07 on brain function and symptoms of AD. These will include:

   o Cognitive Testing:
   * Standard tests like the AD Assessment Scale-Cognitive Subscale (ADAS-cog) and the Mini-Mental State Examination (MMSE) will be used to evaluate any changes in cognitive function.

     o Brain Imaging:
   * MRI scans will help assess changes in brain structure and inflammation.

     o Biomarkers:
   * Blood and CSF samples will be analyzed for specific biomarkers related to inflammation, brain health, and AD progression.
7. Eligibility Criteria

   * Inclusion Criteria:

     * Individuals aged 65-88 with a confirmed diagnosis of MCI or mild to moderate AD.
     * Must have a caregiver who can assist with the study requirements.
     * Must be able to undergo specific procedures like MRI scans and CSF sampling.
   * Exclusion Criteria:

     * Individuals with other significant health conditions or history of neurological disorders other than AD.
     * Those currently participating in another clinical trial or have certain medication restrictions.
8. Importance of the Study AD is a progressive condition that affects memory, thinking, and behavior. Current treatments only manage symptoms temporarily, and there is an need for new therapies. NTRX-07 is a novel drug that has shown promise in animal studies, potentially reducing brain inflammation, clearing harmful proteins, and improving memory and learning. This study is an essential step toward understanding if NTRX-07 can offer a safe and effective treatment option for people with AD.
9. Summary This clinical trial is designed to test the safety and processing of a new drug, NTRX-07, in people with MCI or mild to moderate AD. Participants will be carefully monitored for any side effects while researchers also gather data on the drug's impact on brain function. If successful, this study could lead to more advanced trials and, ultimately, a new treatment option for those affected by AD.

ELIGIBILITY:
Inclusion Criteria

1. Participants must be 65-80 years of age inclusive, at the time of signing the informed consent.
2. Clinical Dementia Rating (CDR) of 0.5 - 2.0; and education-adjusted Logical Memory II scores consistent with MCI or mild to moderate AD (<1.5 SD below mean cutoff). MMSE 12-26
3. pTau 217 consistent with AD, or recent amyloid test panel within 2 years. The test must be after any previous participation in an anti-amyloid MAB trial.
4. Participants who have been in a previous amyloid-directed MAB study must have a negative ARIA report after the study.
5. Confirmed medical documentation of AD symptoms onset at age 60 or later.
6. No active depression and a Geriatric Depression Score of < 6.
7. No change in acetylcholinesterase inhibitors or memantine for the previous six months and is not expected to start an acetylcholinesterase inhibitor during the duration of the study.
8. Living at home, with a reliable caregiver who sees them at least 3 times/week for 10 hours or more and can oversee the administration of the study drug.
9. Provide written informed consent and willingness as documented by a signed informed consent form; responsible caregiver must also provide written consent.
10. Body weight within 55-110 kg and body mass index (BMI) within the range 18-35 kg/m2 (inclusive)
11. Male or Female • Male participants: Male participants are eligible to participate if they agree to the following during the intervention period and for at least 90 days, after the last dose of study intervention:

Refrain from donating sperm PLUS, either:

Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent ba sis) and agree to remain abstinent.

OR

* Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person.

  * Female participants: Must be a woman of nonchildbearing potential (WONCBP) (at least two years post-menopause or surgically sterile).

Exclusion Criteria

1. Reported history or presence of clinically significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data. Participants with stable, well-controlled conditions may be accepted upon review by the investigator and sponsor.
2. Change of more than 2 points from screening MMSE to baseline MMSE, or discrepancy in disease classification between MMSE, and Trail Making test.
3. Diagnosis of a dementia-related CNS disease other than AD (eg, Parkinson's Disease, Huntington's Disease, frontotemporal dementia, multi-infarct dementia, dementia with Lewy bodies, normal pressure hydrocephalus)
4. Cannot tolerate spinal puncture procedure for cerebral spinal fluid (CSF).
5. Anticoagulation therapy that would contraindicate spinal puncture procedure for cerebral spinal fluid (CSF).
6. Any contraindication to MRI (per facility standard of care).
7. Major structural brain disease by reported history or chart review (e.g., ischemic infarcts, subdural hematoma, hemorrhage, hydrocephalus, brain tumors, multiple subcortical ischemic lesions, severe mi- microangiopathic disease, volume loss disproportionate for age or a single lesion in a critical region e.g., thalamus, hippocampus).
8. Findings on MRI demonstrating intracranial pathology as an alternative cause for cognitive impairment
9. Any other reported history of central nervous system (CNS) trauma (e.g., contusion), or infections (e.g., human immunodeficiency virus [HIV], syphilis), that present active or residual effects on cognitive function.
10. Reported history of seizures, with the exception of childhood febrile seizures or metabolic seizures where the underlying etiology has resolved, and the participant has been seizure-free without treatment for at least 2 years.
11. Autoimmune disorders, active infections or other disorders, including the use of immunosuppressants, that may affect the subject's immune system.
12. Reported current or chronic history of clinically significant liver disease. This includes but is not limited to hepatitis virus infections, drug- or alcohol-related liver disease, nonalcoholic steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, or any other liver disease considered clinically significant by the investigator.
13. Reported hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) that are deemed clinically significant by the PI or medical monitor.
14. Abnormal TSH, fT3 or fT4 at baseline screening. Subjects with known hypothyroidism or hyperthyroidism should be stable on treatment for 6 months prior to starting study and not anticipated to require any type of dose adjustment during the course of the study.
15. Reside in a nursing home or assisted care facility with the need for direct continuous medical care and nursing supervision. Participant may reside in such facilities provided continuous direct medical care is not required.
16. Subjects who require close or continual monitoring for self care or basic activities of daily living.
17. Subjects with history of psychiatric conditions such as schizophrenia and or bipolar disorder
18. Any reported history from the patient, family, or on supplied chart re- view or current suicide risk
19. Patients may continue prior concomitant medications at the same sta ble dose. Drugs with potential interactions are detailed in the investi gator's brochure. Participants receiving drugs with strong interactions should be excluded where the drug in question cannot be safely stopped for an appropriate washout period pre-study and until 7 days after the last dose of study medication (completion of the post-study safety visit).
20. Reported treatment with biological agents in the 3 months prior to dosing in this study, or within 5 half-lives of the biological agent prior to dosing..
21. Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investiga- tional study intervention.
22. Clinical laboratory findings outside the normal range and determined by the investigator or medical monitor to be clinically significant. These include but are not limited to:

    1. Alanine transaminase (ALT) or aspartate transaminase (AST) >1.5 x upper limit of normal (ULN)
    2. Total bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35%)
    3. QTcF >450 msec for male participants or >470 msec for female participants
    4. Positive drug/alcohol screen
23. Reported sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study
24. Reported regular use of known drugs of abuse within the past 3 years.
25. Inability to withhold CNS medications (e.g., benzodiazepines, stimulants) for 3 half-lives of the drug prior to cognitive testing and EEG administration.
26. Presence of any contraindication to venous blood sampling for pharmacokinetic analyses.
27. Positive SARS-CoV-2 test, hepatitis panel (including hepatitis B sur face antigen [HBsAg] or hepatitis C virus antibody [anti-HCV]), a positive HIV antibody screen or positive syphilis test

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event incidence in NTRX-07 treated participants | From date of randomization through final study visit, up to 6 weeks.
  Incidence of adverse events during the trial, compared between the active treatment and placebo groups, through study completion, about 6 weeks.

SECONDARY OUTCOMES:
Plasma Pharmacokinetics of NTRX-07 - Area under the curve | First day of dosing and Day 28
  Mean area under the curve determined by plasma levels from time zero to 10 hrs post-dose
Plasma Pharmacokinetics of NTRX-07 - Maximum concentration | First day of dosing and Day 28
  Mean Maximum concentration determined by plasma levels from time zero to to 10 hrs post-dose
Cerebrospinal fluid Pharmacokinetics of NTRX-07 - concentration compared to simultaneous plasma levels | Day 28
  Mean ratio of CSF concentration to plasma levels at 90 minutes post-dose
Change in ADAS-cog in treated participants from baseline | Baseline and Day 28
Change in MMSE in treated participants from baseline | Baseline and day 28.
Change in Free-water by MRI in treated participants | Baseline and last day of dosing + up to 5 days
  Free water determined by MRI as a measure of neuroinflammation
Change in Cortical Disarray Measurement (CDM) determined by MRI in treated subjects | Baseline and last day of dosing + up to 5 days
  Cortical Disarray Measurement as measure of neuronal interconnectivity
Change in Quantitative EEG in treated participants | Baseline and Day 28
  32 lead EEG; absolute power and relative power in the different frequency bands, 10 min eyes shut followed by 10 min eyes open. EEG processing involves the computation of the spectra of artifact-free segments. The Hanning window is used, and the FFT algorithm is analyzed using Matlab scripts. The AUC of spectrum segments provides estimations of power in each frequency band of interest. Absolute powers and relative powers are provided for each band. For each band, relative power is the absolute power divided by the power of the total band.
Change in Quantitative EEG p-300 evoked response in treated participants | Baseline and Day 28
  The P300 wave is an evoked potential that reflects the decision-making process in the cerebral cortex in a situation of cognitive task. It is obtained by repeated stimulations with two types of auditory stimuli: a group of stimuli constituting the background (stimuli called "standard" or "frequent"), against different stimuli which are less frequent (stimuli named "odd" or "rare" or "deviant"). The P300 wave is characterized by a positive deflection occurring approximately 300 ms after odd stimuli.
  The standard stimulus is a 500Hz sound, and the oddball stimulus is a 2000Hz sound. Stimuli are presented through calibrated headphone in a pseudo randomized order. The inter-stimulus interval is randomized between 1200 and 1900ms to avoid anticipation. Oddball makes up 15% of presentations.
Change in Plasma biomarkers in treated participants | Baseline and Day 28
  High-sensitivity C-Reactive Protein (hsCRP), HbA1, erythrocyte sedimentation rate (ESR), TNF-a, IL-1b, IL-6, IL-2, YKL- 40, sTREM2, Abeta40, Abeta42, ptau217
Change in CSF biomarkers in treated participants | Baseline and Day 28
  TNF-a, IL-1b, IL-6, IL-2, YKL- 40, sTREM2, Abeta40, Abeta42, ptau217, Neurogranin, synaptotagmin-1, NfL, GFAP

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Foss, MD, Study Director — NeuroTherapia, Inc.
Locations (5):
- Czechia (2):
  - Neuro Health Centrum s.r.o., Brno
  - Neuropsychiatrie s.r.o., Prague
- Semmelweis University, Budapest, Hungary
- Poland (2):
  - Szpital Uniwersytecki W Krakowie, Krakow
  - Wrocławskie Centrum Alzheimerowskie, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
To be determined. Key elements of safety and biomarker endpoints will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12 months after study closure and publication in a peer-reviewed journal. Information will be maintained for at least 3 years.
Access Criteria: A central publically available repository will be used. The repository will manage data access and permissions. Individual data points with a limited set of patient identifiers will be provided. GDPR regulations will be observed.